CLINICAL TRIAL: NCT00248742
Title: The Impact of Psychobiological Factors in Inflammatory Bowel Disease
Brief Title: Psychobiology in Inflammatory Bowel Disease(IBD)
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Aker (Other); Haukeland University Hospital (Other); University of Bergen (Other); Lübeck University Clinic (Other); University Hospital, Akershus (Other)
Responsible Party: Birgitte Boye MD PhD, Rikshsoptialet University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-00093; 2005/188-2 FBB/-
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-03

CONDITIONS: Inflammatory Bowel Disease
Keywords: IBD, psychological, stress management
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Psychological behavioral intervention — 3x3 hours group intervention followed by 6-9 hours individual psychotherapy based on cognitive behavioral methods
  Other Names: stress management

SUMMARY:
Patients with ulcerous colitis and Crohn's disease, age 18-60, with a relapse within the last 18 months and an activity index ≥4, with a long time stress level ≥60 on the perceived stress questionnaire (PSQ) were randomized to a stress management intervention program or treatment as usual and followed up for 18 months.

DETAILED DESCRIPTION:
The study includes distressed patients with ulcerous colitis and Crohn's disease with relapse or enduring activity last 18 months and an simple activity index ≥4, on stable medication last 4 weeks. All patients were followed by a gastroenterologist at baseline, 3, 6, 12 and 18 months follow up and a psychiatrist or clinical psychologist at 18 months. Half of the patients received additional psychosocial intervention (education, relaxation, supportive psychotherapy with stress management). Assessments include gastrointestinal assessments; blood tests; psychiatric evaluations and psychometric evaluations.

ELIGIBILITY:
Ulcerous colitis and Crohn's disease verified by histology and endoscope Relapse last 18 months or enduring activity Activity index≥4 PSQ≥60

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2001-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Improvement in activity index. | 18 months

SECONDARY OUTCOMES:
Reduction of inflammatory parameters. | 18 months
Reduction in number of relapses. | 18 months
Quality of life improvement | 18 months
Psychobiological factors related to improvement | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Georg Høyer, MD, Study Director — Psychological behavioral intervention based on cognitive behavioral methods
Locations (1):
- RRHF, Oslo, Norway

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391